CLINICAL TRIAL: NCT02296255
Title: Effective Surveillance and Impact of HPV Vaccination on Screening for Cervical Cancer in Tuscany
Brief Title: Effect of HPV Vaccination on Women Aged 25 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cancer Prevention and Research Institute, Italy (Other)
Collaborators: Istituto Toscano Tumori (Other); University of Florence (Other)
Responsible Party: Principal Investigator, Francesca Carozzi, Biologist Director, Cancer Prevention and Research Institute, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F11J09000350002; 342/2009 (Other: Local Ethics Committee of Local Health Unit of Florence)
Record Dates: First submitted 2014-11-11; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Cervical Cancer
Keywords: cervical cancer screening; young women vaccination; impact of HPV vaccination on screening
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no HPV vaccine (No Intervention): No delivery of HPV vaccine
- HPV vaccine (Cervarix®, GlaxoSmithKline) (Experimental): Delivery of HPV vaccine (Cervarix®, GlaxoSmithKline) at 0, 1, 6 months
  Interventions: Biological: Cervarix®, GlaxoSmithKline

INTERVENTIONS:
Biological: Cervarix®, GlaxoSmithKline — 3 doses (0,1,6 months) of Cervarix®, GlaxoSmithKline
  Arms: HPV vaccine (Cervarix®, GlaxoSmithKline)

SUMMARY:
The purposes of this study are to evaluate the effectiveness of vaccination in 25-year old women at the time of their first access to cervical cancer screening, to understand the impact of vaccination on screening activity; to evaluate the immune response following vaccination; to study the dynamics of the infection after vaccination, including the possible change in the frequency of non-vaccine HPV types, to evaluate cytological abnormalities reductions in vaccinated women and to assess if HPV test in urine sample could be a useful non-invasive method to monitor HPV status in younger women.

DETAILED DESCRIPTION:
The present trial, funded by Istituto Toscano Tumori, started in 2010 and was directed to all women aged 25 (birth cohorts 1985 and 1986), resident in the province of Florence and targeted by the screening program. After receiving approval from the Ethics Committee of the Local Health Unit of Florence, women were invited by invitation letter containing a clear description of the study. All women complying with the invitation were asked to fill in the informed consent document.

Women were randomized 1:2 in the Experimental Arm or in the Control Arm. At enrollment, women in the Experimental Arm, after collection of cervical samples (for Pap-test and HPV test), blood sample (for HPV antibody testing on serum before vaccination) and one first void urine sample (for HPV testing), received free vaccination with Cervarix® (vaccine against HPV 16 and 18, 3 doses scheduled). Women in the Control Arm received usual care, i.e. the collection of cervical sample for Pap test.

All women who signed the informed consent have been enrolled regardless of being sexually active or not. For virgo women cervical sample was not collected.

At the second round of screening (30 months since enrollment), women in both Arms were asked to collect cervical samples (for Pap-test and HPV test) while a new blood sample for HPV antibody testing was collected only in women enrolled in the Experimental Arm.

Women with normal cytology in Control Arm and women with HPV-negative result and normal cytology in Experimental Arm, received a recommendation by mail to repeat screening test after 3 years. Women with abnormal Pap test (Atypical Squamous Cells of Undetermined Significance or more severe, ASC-US+) were referred to immediate colposcopy at the Cancer Prevention and Research Insitute. Women with normal cytology and HPV positive were called after one year to repeat HPV test and Pap test. If HPV and Pap test were negative, women repeated both test after 30 months from enrolment. Otherwise if HPV test remained positive and/or cytology abnormalities were detected women were referred for colposcopy: if colposcopy didn't reveal high grade lesions (≤ CIN2) women repeated HPV and Pap test after 30 months from enrollment, if colposcopy revealed final histological diagnosis of CIN2+ lesions, women were recommended for an excisional treatment (both for study and control group).

The presence of high risk (HR) HPVs was evaluated by Hybrid Capture 2 (Qiagen, Gaithersburg, USA) using probe B for the detection of 12 high risk HPV types: 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59 (Group 1) and 1 "probably carcinogenic to humans" type HPV 68 (Group 2).

HPV genotyping was performed by INNO-LiPA Genotyping Extra that allows the identification of 28 different HPV types on L1 region on the HPV genome, it identifies all known HPV high-risk types (Group 1) 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59; "probably carcinogenic to humans" (Group 2A) HPV68; and all "possibly carcinogenic" HPV 26, 53, 66, 69, 70, 73, 82 (Group 2B) and "not classified as to its carcinogenicity to humans" (Group 3) (6, 11); and other HPV types: 40, 43, 44, 54, 71, 74.

HPV antibody testing was performed on an established and validated HPV serology method based on Luminex technology heparin coating of the beads and pseudovirions (PsVs) of 17 HPV types belonging to alpha species: 3, 6, 11, 16, 18, 31, 32 ,33, 35, 39, 45, 52, 56, 58, 59, 68, 73, and for four HPV types belonging to beta species: 5, 15, 38, 76.

ELIGIBILITY:
Inclusion Criteria:

* resident in Florence
* invited for the first time to the cervical cancer screening in Florence
* aged 25 years

Exclusion Criteria:

-

Ages: 25 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 832 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
number of HR-HPV infections and number of infections due to HPV vaccine types in cervical sample in the Experimental arm and in No intervention arm | 30 months
number of cytological abnormalities in the Experimental arm and in No intervention arm | 30 months

SECONDARY OUTCOMES:
Number of subjects seropositive for HPV 16, 18, 31, 33, 35, 39, 45, 52, 56, 58, 59, 68 at enrollment | enrollment
Number of subjects seropositive for HPV16,18 31, 33, 35, 39, 45, 52, 56, 58, 59, 68 after vaccination | 30 months
Anti-HPV16,18 31, 33, 35, 39, 45, 52, 56, 58, 59, 68 Antibody Titers before vaccination | at enrollment
  Titers are given as Mean Fluorescence Intensity Unit (MFI)
Anti-HPV16,18 31, 33, 35, 39, 45, 52, 56, 58, 59, 68 Antibody Titers after vaccination | 30 months
  Titers are given as Mean Fluorescence Intensity Unit (MFI)
Number of participants reporting Adverse Events | within 14 days following any injection
  Adverse Events assessed include Local pain, Local swelling, Local pruritus, Local Erythema, Fever, and every adverse event reported day by day in a diary
HPV identification in urine samples | at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Francesca M Carozzi, PhD, Principal Investigator — Cancer Prevention and Research Institute
Locations (1):
- Cancer Prevention and Research Institute, ISPO, Florence, FI, Italy

REFERENCES:
- [Result] Levi M, Bonanni P, Burroni E, Bechini A, Boccalini S, Sani C, Bonaiuti R, Indiani L, Azzari C, Lippi F, Carozzi F; HPV Screevacc Working Group. Evaluation of bivalent human papillomavirus (HPV) vaccine safety and tolerability in a sample of 25 year old Tuscan women. Hum Vaccin Immunother. 2013 Jul;9(7):1407-12. doi: 10.4161/hv.24337. Epub 2013 Apr 9. PMID 23571176
- [Result] Burroni E, Bonanni P, Sani C, Lastrucci V, Carozzi F; Hpv ScreeVacc Working Group; Iossa A, Andersson KL, Brandigi L, Di Pierro C, Confortini M, Levi M, Boccalini S, Indiani L, Sala A, Tanini T, Bechini A, Azzari C. Human papillomavirus prevalence in paired urine and cervical samples in women invited for cervical cancer screening. J Med Virol. 2015 Mar;87(3):508-15. doi: 10.1002/jmv.24085. Epub 2014 Nov 21. PMID 25418873
- [Derived] Carozzi FM, Ocello C, Burroni E, Faust H, Zappa M, Paci E, Iossa A, Bonanni P, Confortini M, Sani C. Effectiveness of HPV vaccination in women reaching screening age in Italy. J Clin Virol. 2016 Nov;84:74-81. doi: 10.1016/j.jcv.2016.09.011. Epub 2016 Oct 3. PMID 27728850